CLINICAL TRIAL: NCT03945344
Title: Effect of Charcoal on Gastrointestinal Absorption of Tiotropium; A Randomised, Open, Single Centre, Single Dose, Crossover Study in Healthy Subjects
Brief Title: Effect of Charcoal on Gastrointestinal Absorption of Tiotropium
Acronym: TIOBLOCK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3122003
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Tiotropium with concomitant charcoal
  Interventions: Drug: Tiotropium
- Treatment B (Experimental): Tiotropium without concomitant charcoal.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium — Oral capsule 20 μg
  Arms: Treatment A
Drug: Tiotropium — Oral capsule 20 μg
  Arms: Treatment B

SUMMARY:
The study will assess how efficiently activated charcoal will block absorption of tiotropium via the gastro intestinal track. Pharmacokinetics of tiotropium will be compared after orally administered tiotropium capsule with and without concomitant activated charcoal administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Healthy males and females, aged 18-60
3. Normal weight at least 50 kg.

Exclusion Criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological or psychiatric disease.
2. Any condition requiring regular concomitant treatment (including vitamins and herbal products) or likely to need any concomitant treatment during the study.
3. Any clinically significant abnormal laboratory value or physical finding that may interfere the interpretation of study result or constitute a health risk for the subject if he/she participates in the study.
4. Known hypersensitivity to tiotropium bromide, atropine or its derivatives or to the excipients of the drug.
5. Pregnant or lactating females.
6. Females of childbearing potential not using proper contraception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameter Area Under Curve (AUC) | 24 hours

SECONDARY OUTCOMES:
Peak concentration in plasma (Cmax) and time to reach peak concentration in plasma (tmax) | (0 hours) and at 15, 30 and 45 minutes, and 1,1.5, 2, 3, 3.5, 4, 4.5, 5, 6, 8, 12 and 24 hours after the administration

CONTACTS AND LOCATIONS:
Overall Officials: Maria Annunen, MSc, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Clinical Pharmacology Unit, Espoo, Finland